CLINICAL TRIAL: NCT04147156
Title: Efficacy of a New Type of Mechanical Rotational Chair (ROTUNDUM) in Treating BPPV
Brief Title: Efficacy of a New Type of Mechanical Rotational Chair in Treating BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dan Dupont Hougaard, MD, Associate Professor, Principal Investigator, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROTDUNDUM1
Record Dates: First submitted 2019-10-30; First posted 2019-10-31 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: BPPV
Keywords: Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular diseases; Epley Maneuver; Semont Maneuver; Repositioning chair
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo; Vertigo; Dizziness; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epley's Maneuver (Active Comparator): Treatment of posterior canal BPPV with Epley's maneuver in the ROTUNDUM-chair.
  Interventions: Procedure: Epley's Maneuver
- Semont Maneuver (Experimental): Treatment of posterior canal BPPV with the Semont maneuver in the ROTUNDUM-chair.
  Interventions: Procedure: Semont Maneuver
- 360 degree vertical rotation (Active Comparator): Treatment of posterior canal BPPV with a 360 degree vertical rotation in the ROTUNDUM-chair.
  Interventions: Procedure: 360 degree vertical rotation

INTERVENTIONS:
Procedure: Epley's Maneuver — Treatment with Epley's Maneuver in the ROTUNDUM-chair
  Arms: Epley's Maneuver
Procedure: Semont Maneuver — Treatment with the Semont Maneuver in the ROTUNDUM-chair
  Arms: Semont Maneuver
Procedure: 360 degree vertical rotation — Treatment with 360 degree vertical rotation in the ROTUNDUM-chair
  Arms: 360 degree vertical rotation

SUMMARY:
A study to establish the efficacy of a new type of mechanical rotational chair in treating BPPV. In addition, comparison of three types of treatment maneuvers using the mechanical rotational chair.

DETAILED DESCRIPTION:
Open-label, randomized controlled trial comparing three different treatment maneuvers in a mechanical rotational chair (ROTUNDUM-chair) in treating BPPV. Patients diagnosed with BPPV will be randomized to one of three maneuvers in the ROTUNDUM-chair:

1. Epley's maneuver
2. Semont maneuver
3. 360 degree vertical rotation

ELIGIBILITY:
Inclusion Criteria:

* Characteristic (for BPPV) positional nystagmus
* Positive Dix-Hallpike Test
* Medical history compatible with BPPV

Exclusion Criteria:

* Treatment in a mechanical rotational chair within the last 6 months
* Exclusion of BPPV diagnosis
* Lack of treatment cooperation
* Known cerebral aneurism or cerebral hemorrhage
* Treated for BPPV within the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Number of treatments | 2 years
  Number of treatments necessary to achieve resolution of vertigo and nystagmus
Treatment success after first treatment | 2 years
  Number of subjects achieving resolution of vertigo and nystagmus after one treatment

SECONDARY OUTCOMES:
Dizziness Handicap Inventory (DHI) questionnaire | 2 years
  Comparison of pre- and post-treatment score, total score between 0 and 100. Higher score reflects worse condition
Adverse events | 2 years
  Registration of adverse events
Value of liberatory nystagmus | 2 years
  Registration of liberatory nystagmus after each treatment as a prognostic factor for treatment success

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Hougaard, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No